CLINICAL TRIAL: NCT02011360
Title: Evidence-Based Approach to Dietary Management of Prader-Willi Syndrome (PWS)
Brief Title: Prader-Willi Syndrome Macronutrient Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Foundation for Prader-Willi Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: Pro00049226; SFR2382 (Other Grant/Funding Number: Foundation for Prader-Willi Research (US))
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Prader Willi Syndrome; Syndromic Obesity; Childhood Obesity
Keywords: Prader Willi syndrome; childhood obesity; ghrelin; appetite regulation
MeSH Terms: conditions — Prader-Willi Syndrome; Pediatric Obesity | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

ARMS (2):
- Low carbohydrate diet (Other): Low carbohydrate diet: 15%carb; 65%fat; 20% protein. This will be administered over 72 hour hospital stay.
  Interventions: Other: Low Fat diet
- Low Fat diet (Other): Low fat diet: 65%carb; 15%fat; 20% protein. This will be administered over a 72 hour hospital stay.
  Interventions: Other: Low Carbohydrate diet

INTERVENTIONS:
Other: Low Carbohydrate diet — Low carbohydrate diet: 15%carb; 65%fat; 20% protein
  Arms: Low Fat diet
Other: Low Fat diet — Low Fat diet: 65%carb; 15%fat; 20% protein
  Arms: Low carbohydrate diet

SUMMARY:
The overall objective is to explore the mechanisms by which macronutrients regulate food intake and weight gain in Prader Willi Syndrome (PWS).

Previous studies from the investigators' labs suggest that the increased appetite of PWS may be triggered or maintained by an increase in the levels of ghrelin, an appetite-stimulating hormone produced primarily by the stomach. This study will compare the effects of low carbohydrate diet versus low fat diet on levels of ghrelin, appetite suppressing hormones and markers of insulin sensitivity in patients with PWS.

The investigators hypothesize that the low carbohydrate diet will suppress plasma active ghrelin and increase appetite-suppressing hormones to a greater degree and for longer duration than the low fat diet and will thereby reduce hyperphagia and increase satiety. The investigators also hypothesize that the low carb diet will improve hormonal and metabolic markers (fatty acids, amino acids and organic acids) of insulin sensitivity and inflammatory cytokine profiles of children with PWS.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Prader Willi syndrome confirmed by chromosome analysis (ie. interstitial deletion of paternally-derived chromosome 15q, uniparental maternal disomy or other chromosome 15 abnormalities)
* age 5 years to 17 years
* written informed consent and assent obtained and willingness to comply with the study schedule and procedures
* free T4, TSH values in the normal range (either endogenous or with thyroxine replacement)
* weight stable (BMI percentile fluctuation of <5 percentiles) over the preceding 2 months prior to the study

Exclusion Criteria:

* presence of other clinically significant disease that would impact body composition including diabetes mellitus, chronic inflammatory bowel disease, chronic severe liver or kidney disease or neurologic disorders
* concomitant use of medications known to affect body weight or investigational drug in the past year

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Suppression of ghrelin | 10 hour fast following completion of dietary intervention
  Fasting labs will be obtained immediately following dietary intervention. These labs will include total and active ghrelin.

SECONDARY OUTCOMES:
Changes in satiety | During the 72 hour dietary intervention
  Changes in subjective hunger will be assessed by an appetite and hyperphagia questionnaire validated for PWS children. This will be completed by the children, with assistance of their parents, at completion of the 72 hour dietary intervention.
Improvements in insulin sensitivity | During the 72 hour dietary intervention.
  The analysis will include measurements of adiponectin, GLP-1, glucose, insulin, AST, ALT, insulin sensitivity and a detailed profile ("metabolomics") of amino acids, fatty acids, acylcarnitines, and adipocytokines on the day prior to and immediately following dietary intervention.

OTHER OUTCOMES:
Improvement in inflammatory cytokine profile | During the 72 hour dietary intervention
  The analysis will include measurements of adiponectin, GLP-1, glucose, insulin, AST, ALT, insulin sensitivity and a detailed profile ("metabolomics") of amino acids, fatty acids, acylcarnitines, and adipocytokines on the day prior to and immediately following dietary intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Freemark, MD, Principal Investigator — Duke University; Andrea M Haqq, MD, Principal Investigator — University of Alberta
Locations (2):
- Duke University Medical Center, Durham, North Carolina, United States
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Dykens EM, Maxwell MA, Pantino E, Kossler R, Roof E. Assessment of hyperphagia in Prader-Willi syndrome. Obesity (Silver Spring). 2007 Jul;15(7):1816-26. doi: 10.1038/oby.2007.216. PMID 17636101
- [Background] Haqq AM, Muehlbauer M, Svetkey LP, Newgard CB, Purnell JQ, Grambow SC, Freemark MS. Altered distribution of adiponectin isoforms in children with Prader-Willi syndrome (PWS): association with insulin sensitivity and circulating satiety peptide hormones. Clin Endocrinol (Oxf). 2007 Dec;67(6):944-51. doi: 10.1111/j.1365-2265.2007.02991.x. Epub 2007 Jul 30. PMID 17666087
- [Background] Haqq AM, Muehlbauer MJ, Newgard CB, Grambow S, Freemark M. The metabolic phenotype of Prader-Willi syndrome (PWS) in childhood: heightened insulin sensitivity relative to body mass index. J Clin Endocrinol Metab. 2011 Jan;96(1):E225-32. doi: 10.1210/jc.2010-1733. Epub 2010 Oct 20. PMID 20962018
- [Background] Haqq AM, Farooqi IS, O'Rahilly S, Stadler DD, Rosenfeld RG, Pratt KL, LaFranchi SH, Purnell JQ. Serum ghrelin levels are inversely correlated with body mass index, age, and insulin concentrations in normal children and are markedly increased in Prader-Willi syndrome. J Clin Endocrinol Metab. 2003 Jan;88(1):174-8. doi: 10.1210/jc.2002-021052. PMID 12519848
- [Background] Cummings DE, Clement K, Purnell JQ, Vaisse C, Foster KE, Frayo RS, Schwartz MW, Basdevant A, Weigle DS. Elevated plasma ghrelin levels in Prader Willi syndrome. Nat Med. 2002 Jul;8(7):643-4. doi: 10.1038/nm0702-643. No abstract available. PMID 12091883
- [Background] Haqq AM, Grambow SC, Muehlbauer M, Newgard CB, Svetkey LP, Carrel AL, Yanovski JA, Purnell JQ, Freemark M. Ghrelin concentrations in Prader-Willi syndrome (PWS) infants and children: changes during development. Clin Endocrinol (Oxf). 2008 Dec;69(6):911-20. doi: 10.1111/j.1365-2265.2008.03385.x. Epub 2008 Aug 15. PMID 18710462
- [Background] Newgard CB, An J, Bain JR, Muehlbauer MJ, Stevens RD, Lien LF, Haqq AM, Shah SH, Arlotto M, Slentz CA, Rochon J, Gallup D, Ilkayeva O, Wenner BR, Yancy WS Jr, Eisenson H, Musante G, Surwit RS, Millington DS, Butler MD, Svetkey LP. A branched-chain amino acid-related metabolic signature that differentiates obese and lean humans and contributes to insulin resistance. Cell Metab. 2009 Apr;9(4):311-26. doi: 10.1016/j.cmet.2009.02.002. PMID 19356713
- [Background] Laferrere B, Reilly D, Arias S, Swerdlow N, Gorroochurn P, Bawa B, Bose M, Teixeira J, Stevens RD, Wenner BR, Bain JR, Muehlbauer MJ, Haqq A, Lien L, Shah SH, Svetkey LP, Newgard CB. Differential metabolic impact of gastric bypass surgery versus dietary intervention in obese diabetic subjects despite identical weight loss. Sci Transl Med. 2011 Apr 27;3(80):80re2. doi: 10.1126/scitranslmed.3002043. PMID 21525399
- [Background] Wang TJ, Larson MG, Vasan RS, Cheng S, Rhee EP, McCabe E, Lewis GD, Fox CS, Jacques PF, Fernandez C, O'Donnell CJ, Carr SA, Mootha VK, Florez JC, Souza A, Melander O, Clish CB, Gerszten RE. Metabolite profiles and the risk of developing diabetes. Nat Med. 2011 Apr;17(4):448-53. doi: 10.1038/nm.2307. Epub 2011 Mar 20. PMID 21423183
- [Background] Sondike SB, Copperman N, Jacobson MS. Effects of a low-carbohydrate diet on weight loss and cardiovascular risk factor in overweight adolescents. J Pediatr. 2003 Mar;142(3):253-8. doi: 10.1067/mpd.2003.4. PMID 12640371
- [Background] Foster GD, Wyatt HR, Hill JO, McGuckin BG, Brill C, Mohammed BS, Szapary PO, Rader DJ, Edman JS, Klein S. A randomized trial of a low-carbohydrate diet for obesity. N Engl J Med. 2003 May 22;348(21):2082-90. doi: 10.1056/NEJMoa022207. PMID 12761365
- [Background] Samaha FF, Iqbal N, Seshadri P, Chicano KL, Daily DA, McGrory J, Williams T, Williams M, Gracely EJ, Stern L. A low-carbohydrate as compared with a low-fat diet in severe obesity. N Engl J Med. 2003 May 22;348(21):2074-81. doi: 10.1056/NEJMoa022637. PMID 12761364
- [Background] Stern L, Iqbal N, Seshadri P, Chicano KL, Daily DA, McGrory J, Williams M, Gracely EJ, Samaha FF. The effects of low-carbohydrate versus conventional weight loss diets in severely obese adults: one-year follow-up of a randomized trial. Ann Intern Med. 2004 May 18;140(10):778-85. doi: 10.7326/0003-4819-140-10-200405180-00007. PMID 15148064
- [Background] Brehm BJ, Seeley RJ, Daniels SR, D'Alessio DA. A randomized trial comparing a very low carbohydrate diet and a calorie-restricted low fat diet on body weight and cardiovascular risk factors in healthy women. J Clin Endocrinol Metab. 2003 Apr;88(4):1617-23. doi: 10.1210/jc.2002-021480. PMID 12679447
- [Background] Yancy WS Jr, Olsen MK, Guyton JR, Bakst RP, Westman EC. A low-carbohydrate, ketogenic diet versus a low-fat diet to treat obesity and hyperlipidemia: a randomized, controlled trial. Ann Intern Med. 2004 May 18;140(10):769-77. doi: 10.7326/0003-4819-140-10-200405180-00006. PMID 15148063
- [Background] Dansinger ML, Gleason JA, Griffith JL, Selker HP, Schaefer EJ. Comparison of the Atkins, Ornish, Weight Watchers, and Zone diets for weight loss and heart disease risk reduction: a randomized trial. JAMA. 2005 Jan 5;293(1):43-53. doi: 10.1001/jama.293.1.43. PMID 15632335
- [Background] Bistrian BR, Blackburn GL, Stanbury JB. Metabolic aspects of a protein-sparing modified fast in the dietary management of Prader-Willi obesity. N Engl J Med. 1977 Apr 7;296(14):774-9. doi: 10.1056/NEJM197704072961402. PMID 840278
- [Background] Fields DA, Higgins PB, Radley D. Air-displacement plethysmography: here to stay. Curr Opin Clin Nutr Metab Care. 2005 Nov;8(6):624-9. doi: 10.1097/01.mco.0000171127.44525.07. PMID 16205463
- [Background] Day N, McKeown N, Wong M, Welch A, Bingham S. Epidemiological assessment of diet: a comparison of a 7-day diary with a food frequency questionnaire using urinary markers of nitrogen, potassium and sodium. Int J Epidemiol. 2001 Apr;30(2):309-17. doi: 10.1093/ije/30.2.309. PMID 11369735
- [Background] Stubbs RJ, Hughes DA, Johnstone AM, Rowley E, Reid C, Elia M, Stratton R, Delargy H, King N, Blundell JE. The use of visual analogue scales to assess motivation to eat in human subjects: a review of their reliability and validity with an evaluation of new hand-held computerized systems for temporal tracking of appetite ratings. Br J Nutr. 2000 Oct;84(4):405-15. doi: 10.1017/s0007114500001719. PMID 11103211
- [Background] Liu J, Prudom CE, Nass R, Pezzoli SS, Oliveri MC, Johnson ML, Veldhuis P, Gordon DA, Howard AD, Witcher DR, Geysen HM, Gaylinn BD, Thorner MO. Novel ghrelin assays provide evidence for independent regulation of ghrelin acylation and secretion in healthy young men. J Clin Endocrinol Metab. 2008 May;93(5):1980-7. doi: 10.1210/jc.2007-2235. Epub 2008 Mar 18. PMID 18349056
- [Background] Haqq AM, Lien LF, Boan J, Arlotto M, Slentz CA, Muehlbauer MJ, Rochon J, Gallup D, McMahon RL, Bain JR, Stevens R, Millington D, Butler MD, Newgard CB, Svetkey LP. The Study of the Effects of Diet on Metabolism and Nutrition (STEDMAN) weight loss project: Rationale and design. Contemp Clin Trials. 2005 Dec;26(6):616-25. doi: 10.1016/j.cct.2005.09.003. Epub 2005 Oct 18. PMID 16239128
- [Background] Nass R, Liu J, Hellmann P, Coschigano KT, Gaylinn B, Berryman DE, Kopchick JJ, Thorner MO. Chronic changes in peripheral growth hormone levels do not affect ghrelin stomach mRNA expression and serum ghrelin levels in three transgenic mouse models. J Neuroendocrinol. 2004 Aug;16(8):669-75. doi: 10.1111/j.1365-2826.2004.01220.x. PMID 15271059